CLINICAL TRIAL: NCT00153920
Title: Phase II Trial of Velcade (Bortezomib) in Patients With Previously Untreated Multiple Myeloma
Brief Title: Bortezomib (Velcade) in Patients With Untreated Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Roswell Park Cancer Institute (Other); Emory University (Other); Memorial Sloan Kettering Cancer Center (Other); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Paul G. Richardson, MD, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-328
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Velcade; bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bortezomib (Experimental): Participants received intravenous bortezomib on a 3-week dosing cycle: 1.3 mg/m2 on days 1, 4, 8 and 11 followed by 10 day rest period for up to 8 cycles or for 2 cycles beyond complete response. Participants with progressive disease or unacceptable toxicity discontinued treatment.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib
  Other Names: Velcade

SUMMARY:
Bortezomib (Velcade) has just recently been approved by the FDA for the treatment of multiple myeloma in patients who have received at least two prior therapies and have demonstrated disease progression on the last therapy. This study will determine if Velcade is effective in treating patients with multiple myeloma that have had no prior treatment for the disease. We will also use whole-genome scanning to identify drug response biomarkers in bone marrow samples as well as nerve fiber studies to compare nerves prior to the use of Velcade and after treatment with Velcade.

DETAILED DESCRIPTION:
Primary Objective

• To evaluate the objective response rate (CR + PR) to bortezomib alone in patients with newly diagnosed multiple myeloma.

Secondary Objectives

* To evaluate the tolerability and toxicity.
* To evaluate time to progression.
* To assess the frequency and severity of peripheral neuropathy.
* To evaluate the impact of early intervention with dose modification and explore symptomatic treatment of peripheral neuropathy.

Exploratory Objectives

• To perform pharmacogenomic analysis of molecular markers associated with response or non-response.

Statistical Design A one stage design is used to evaluate ORR. With 60 evaluable participants, if at least 27 objective responses are observed then bortezomib will be considered promising. The probability of concluding the treatment promising is >0.95 with a true ORR of 55% and <0.07 with a true ORR of 35%.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma based upon standard criteria
* Measurable disease, defined as a monoclonal immunoglobulin spike on serum electrophoresis of > 1 g/dl and/or urine monoclonal immunoglobulin spike of > 200mg/24 hours.
* Karnofsky performance status of > 60
* Hemoglobin > 8.0 g/dL
* AST (SGOT) < 3 x ULN
* ALT < 3 x ULN
* Total bilirubin < 2 x ULN
* Is infertile or is practicing an adequate form of contraception
* 18 years of age or older

Exclusion Criteria:

* Prior treatment with systemic chemotherapy
* Plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes
* Plasma cell leukemia
* Calculated or measured creatinine clearance < 30 mL/minute within 14 days of enrollment
* Grade 2 or greater peripheral neuropathy
* Hypersensitivity to bortezomib, boron or mannitol
* Severe hypercalcemia
* HIV positive
* Known active hepatitis B or C
* New York Hospital Association Class III or IV heart failure
* Second malignancy requiring concurrent treatment
* Other serious medical or psychiatric illness
* Pregnant women
* Dialysis dependent patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-12; Primary Completion 2007-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Richardson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Richardson PG, Xie W, Mitsiades C, Chanan-Khan AA, Lonial S, Hassoun H, Avigan DE, Oaklander AL, Kuter DJ, Wen PY, Kesari S, Briemberg HR, Schlossman RL, Munshi NC, Heffner LT, Doss D, Esseltine DL, Weller E, Anderson KC, Amato AA. Single-agent bortezomib in previously untreated multiple myeloma: efficacy, characterization of peripheral neuropathy, and molecular correlations with response and neuropathy. J Clin Oncol. 2009 Jul 20;27(21):3518-25. doi: 10.1200/JCO.2008.18.3087. Epub 2009 Jun 15. PMID 19528374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 participants were enrolled between December 2003 and September 2005.
Period: Overall Study
Arm/Group | Bortezomib
Started | 66
Eligible and Treated | 64
Completed | 36
Not Completed | 30
Not completed — Adverse Event | 9
Not completed — Progressive Disease | 9
Not completed — Physician Decision | 3
Not completed — Lack of Response | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Non-Protocol Therapy | 1
Not completed — Withdrawal of Consent before Trt | 1
Not completed — Progressive Disease before Trt | 1

BASELINE CHARACTERISTICS:
Population: The analysis population is comprised of eligible and treated participants.
Arm/Group | Bortezomib
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 60 [33 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 44
Race/Ethnicity, Customized [Number; unit: participants]
  White | 59
  Non-White | 5
Region of Enrollment [Number; unit: participants]
  United States | 64
ISS Stage [Number; unit: participants] — International Staging System (ISS) Stage I: serum ß2-M < 3.5 mg/L and serum albumin >/= 3.5 g/dL Stage II: Neither stage I nor stage III Stage III: serum ß2-M >/= 5.5 mg/L
  participants
    ISS Stage I | 32
    ISS Stage II | 26
    ISS Stage III | 4
    Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR) Rate
Description: Objective response was defined as complete response (CR) or partial response (PR) according to European Group for Blood and Marrow Transplantation criteria (Blade J et al Br J Haematol 1998). CR required all of the following: Negative immunofixation on the serum and urine at two consecutive times for minimum 6 weeks; Disappearance of soft tissue plasmacytomas for at least 6 weeks; <5% plasma cells in bone marrow on 2 determinations for a minimum of 6 weeks; No increase in the size or number of lytic bone lesions. PR required all the following: ≥50% reduction in the level of the serum monoclonal protein on 2 determinations for minimum 6 weeks; If present, reduction in 24-hour urinary light chain excretion either by ≥90% or to <200 mg on 2 determinations for minimum 6 weeks; ≥50% reduction size of soft tissue plasmacytomas for minimum 6 weeks; No increase in the number or size of lytic bone lesions. Development of a compression fracture does not exclude response in either category.
Time Frame: Response was assessed every two cycles on treatment. Treatment duration in months was a median (range) of 5.1 (0.8-6.1).
Population: The analysis population is comprised of eligible and treated participants.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 64
proportion of participants | 0.41 [0.30 to 0.52]

2. Secondary Outcome: Very Good Partial Response (VGPR) Rate
Description: Very good partial response or better was defined per International Uniform Response criteria (Durie B, Harousseau JL, Miquel JS, et al Leukemia 2006). See CR requirements in primary outcome measure plus if serum and urine M protein were unmeasurable then immunoglobulin free light chain (FLC) must be in a normal ratio of 0.26-1.65 at two consecutive times. VGPR required the following: Serum and urine M-component detectable by immunofixation but not on electrophoresis; >=90% reduction in serum M-component plus urine M-component <100 mg per 24 hours (by SPEP and UPEP); if the serum and urine M protein were unmeasurable then a >90% decrease in the difference between involved and uninvolved FLC levels.
Time Frame: Response was assessed every two cycles on treatment. Treatment duration in months was a median (range) of 5.1 (0.8-6.1).
Population: The analysis population is comprised of eligible and treated participants.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 64
proportion of participants | .17 [.089 to .287]

3. Secondary Outcome: Time to Progression (TTP)
Description: TTP based on the Kaplan-Meier method is defined as the time from start of treatment to documentation of disease progression (PD). Participants without evidence of PD were censored at the latest date of last disease assessment or date of initiation of non-protocol therapy. PD was established based European Group for Blood and Marrow Transplantation criteria (Blade J et al Br J Haematol 1998). PD required 1 or more of the following: >25% increase in serum monoclonal protein with absolute minimum of 0.5 g/dL (confirmed on repeat investigation); >25% increase in 24-hour urinary light chain excretion with minimum absolute increase of 200 mg/24 hrs (confirmed on repeat investigation); >25% increase in bone marrow plasma cells with minimum absolute increase of 10%; Definite increase in size of existing or new soft tissue plasmacytomas and/or lytic lesions; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL not attributable to other cause).
Time Frame: Disease was assessed every two cycles on treatment and every 6 weeks in long-term follow-up. Median follow-up was 29 months.
Population: The analysis population is comprised of eligible and treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib
Number analyzed (Participants) | 64
months | 17.3 [10.6 to 23.0]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS based on the Kaplan-Meier method is defined as the time from study entry to the earliest documentation of disease progression (PD) or death. Participants alive without evidence of PD were censored at the earliest date of last disease assessment or date of initiation of non-protocol therapy. PD was established based European Group for Blood and Marrow Transplantation criteria (Blade J et al Br J Haematol 1998). PD required 1 or more of the following: >25% increase in serum monoclonal protein with absolute minimum of 0.5 g/dL (confirmed on repeat investigation); >25% increase in 24-hour urinary light chain excretion with minimum absolute increase of 200 mg/24 hrs (confirmed on repeat investigation); >25% increase in bone marrow plasma cells with minimum absolute increase of 10%; Definite increase in size of existing soft tissue plasmacytomas and/or lytic lesions or new; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL not attributable to other cause).
Time Frame: Disease was assessed every two cycles on treatment and every 6 weeks in long-term follow-up. Median follow-up was 29 months as of the data analysis.
Population: The analysis population is comprised of eligible and treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib
Number analyzed (Participants) | 64
months | 17.0 [8.6 to 21.5]

5. Secondary Outcome: Number of Participants With Treatment-Emergent Sensory Neuropathy
Description: Number of participants experiencing any grade treatment-emergent sensory neuropathy events based on CTCAEv3 as reported on case report forms.
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. Treatment duration in months was a median (range) of 5.1 (0.8-6.1).
Population: The analysis population is comprised of eligible and treated participants.
Measure: Number; unit: participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 64
participants | 41

6. Secondary Outcome: Number of Participants With Treatment-Emergent Neuropathic Pain
Description: Number of participants experiencing any grade treatment-emergent neuropathic pain events based on CTCAEv3 as reported on case report forms.
Time Frame: as for outcome 5
Population: The analysis population is comprised of eligible and treated participants.
Measure: Number; unit: participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 64
participants | 8

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. Treatment duration in months was a median (range) of 5.1 (0.8-6.1).
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with bortezomib treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with bortezomib treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | Bortezomib
Serious Adverse Events (participants affected / at risk) | 33/64
Other Adverse Events (participants affected / at risk) | 62/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=64)
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Fever w/o neutropenia (General disorders) | 1
Edema limb (General disorders) | 1
Pain-other (General disorders) | 1
Infection-other (Infections and infestations) | 2
Leukocytes (Investigations) | 4
Lymphopenia (Investigations) | 14
Neutrophils (Investigations) | 4
Platelets (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1
Neuropathy-motor (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Neuropathic, pain (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=64)
Tinnitus (Nervous system disorders) | 1
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 1
Encephalopathy (Nervous system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 4
Hematologic-other (Blood and lymphatic system disorders) | 1
Lymphatics-other (Blood and lymphatic system disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Dry eye syndrome (Eye disorders) | 3
Double vision (Eye disorders) | 1
Vision-blurred (Eye disorders) | 3
Tearing (Eye disorders) | 4
Ocular-other (Eye disorders) | 7
Constipation (Gastrointestinal disorders) | 32
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 20
Distention/bloating, abdominal (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 33
Vomiting (Gastrointestinal disorders) | 9
GI-other (Gastrointestinal disorders) | 4
Oral cavity, hemorrhage (Gastrointestinal disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 1
Stomach, pain (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 26
Fever w/o neutropenia (General disorders) | 6
Rigors/chills (General disorders) | 4
Constitutional, other (General disorders) | 3
Edema head and neck (General disorders) | 2
Edema limb (General disorders) | 6
Pain-other (General disorders) | 9
Allergic reaction (Immune system disorders) | 2
Allergy-other (Immune system disorders) | 1
Infection Gr0-2 neut, eye NOS (Infections and infestations) | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 1
Infection-other (Infections and infestations) | 2
Leukocytes (Investigations) | 18
Lymphopenia (Investigations) | 7
Neutrophils (Investigations) | 8
Platelets (Investigations) | 25
Weight gain (Investigations) | 1
Weight loss (Investigations) | 7
Alkaline phosphatase (Investigations) | 1
ALT, SGPT (Investigations) | 3
Amylase (Investigations) | 2
AST, SGOT (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 2
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 11
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 6
Joint, pain (Musculoskeletal and connective tissue disorders) | 3
Muscle, pain (Musculoskeletal and connective tissue disorders) | 5
Taste disturbance (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 8
Neuropathy-motor (Nervous system disorders) | 5
Neuropathy-sensory (Nervous system disorders) | 39
Neurologic-other (Nervous system disorders) | 3
Head/headache (Nervous system disorders) | 9
Neuropathic, pain (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Renal/GU-other (Renal and urinary disorders) | 3
Breast, pain (Reproductive system and breast disorders) | 1
Pelvic, pain (Reproductive system and breast disorders) | 1
Testicle, pain (Reproductive system and breast disorders) | 4
Uterus, pain (Reproductive system and breast disorders) | 1
Erectile impotence (Reproductive system and breast disorders) | 1
Sexual/Reproductive function-Other (Reproductive system and breast disorders) | 2
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Sweating (Skin and subcutaneous tissue disorders) | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 15
Skin-other (Skin and subcutaneous tissue disorders) | 4
Hypotension (Vascular disorders) | 4
Hot flashes (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No